CLINICAL TRIAL: NCT02396147
Title: A Phase 1, Open-Label, Randomized, Three-Way Crossover Study Evaluating the Relative Bioavailability and Effect of Food on TAK-385 Tablet Formulations in Healthy Subjects
Brief Title: Bioavailability and Effect of Food on TAK-385 Tablet Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-385-1010; U1111-1165-3720 (Registry Identifier: WHO)
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: T2-A + T4B-B + T4B-C (Experimental): T2 Formulation Regimen A (T2-A) TAK-385, 120 mg tablet (80 mg + 40 mg tablets), orally, under fasted conditions, T4 Formulation B Regimen B (T4B-B) TAK-385, 120 mg tablet, orally, under fasted conditions, and T4 Formulation B Regimen C (T4B-C) TAK-385, 120 mg tablet, orally, under fed conditions. There were 6 randomized sequences. Study medication was administered as a single dose on Days 1, 11 and 21. There was a 10-day washout period between each dose.
  Interventions: Drug: TAK-385 T2 Formulation; Drug: TAK-385 T4 Formulation B
- Arm 2: T2-A + T4C-D + T4C-E (Experimental): T2 Formulation Regimen A (T2-A) TAK-385, 120 mg tablet (80 mg + 40 mg tablets), orally, under fasted conditions, T4 Formulation C Regimen D (T4C-D) TAK-385, 120 mg tablet, orally, under fasted conditions, and T4 Formulation C Regimen E (T4C-E) TAK-385, 120 mg tablet, orally, under fed conditions. There were 6 randomized sequences. Study medication was administered as a single dose on Days 1, 11 and 21. There was 10-day washout period between each dose.
  Interventions: Drug: TAK-385 T2 Formulation; Drug: TAK-385 T4 Formulation C

INTERVENTIONS:
Drug: TAK-385 T2 Formulation — TAK-385 T2 Formulation tablets
Drug: TAK-385 T4 Formulation B — TAK-385 T4 Formulation B tablets
  Arms: Arm 1: T2-A + T4B-B + T4B-C
Drug: TAK-385 T4 Formulation C — TAK-385 T4 Formulation C tablets
  Arms: Arm 2: T2-A + T4C-D + T4C-E

SUMMARY:
The purpose of this study is to evaluate the oral bioavailability of two new tablet formulations of TAK-385 (T4 Formulation B and T4 Formulation C) under fasted and fed conditions, relative the T2 Formulation tablet; and to estimate the effect of food on the pharmacokinetics (PK) of a single oral dose of the T4 Formulation B tablet and the T4 Formulation C tablet.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-385. In this study, two new formulations of TAK-385 are being evaluated under fasted and fed conditions, relative to a previous formulation of TAK-385, to assess its bioavailability and how it is processed by the body. This study will look at lab results of people who take TAK-385.

The study will enroll approximately 54 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups (Arms). Participants in Arm 1 will receive TAK-385 T2 Formulation 120 mg tablet (80mg + 40mg tablets) under fasted conditions, TAK-385 T4 Formulation B 120 mg tablet under fasted conditions, and TAK-385 T4 Formulation B 120 mg tablet under fed conditions. Participants in Arm 2 will receive TAK-385 T2 Formulation 120 mg tablet (80mg + 40mg tablets) under fasted conditions, TAK-385 T4 Formulation C 120 mg tablet under fasted conditions, and TAK-385 T4 Formulation C 120 mg tablet under fed conditions. Participants in each arm will be randomized to receive study drug in one of 6 treatment sequences. Study medication will be administered as a single dose on Days 1, 11 and 21. There will be a 10-day washout period between each dose.

This single-centre trial will be conducted in the United States. The overall time to participate in this study is 51 days. Participants will make 10 visits to the clinic, including three 4-day periods of confinement to the clinic, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 55 years, inclusive, at the time of consent.
2. Healthy adult male, as determined by a physician evaluation that includes:

   * Medical history (ie, no clinically significant medical conditions requiring ongoing drug therapy).
   * Physical examination.
   * Vital signs.
   * Electrocardiogram (ECG).
   * Laboratory evaluation (hematology, biochemistry, and urinalysis).
   * No acute illness within 30 days before screening that required prescription or over-the-counter (OTC) medicines.
3. Weight ≥ 55 kg and body mass index (BMI) between 18.0 and 32.0 kg/m^2 inclusive, at Screening.
4. Nonsmoker for at least 2 years and does not use nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, or nicotine patch or gum).
5. Male participants, even if surgically sterilized (ie, status postvasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
7. Suitable venous access for the study-required blood sampling.
8. Abstains from behavior that increases susceptibility to contract blood-borne pathogens (eg, obtaining a tattoo or participating in unsafe needle use for any purpose) during the 28 days before study entry.
9. In the opinion of the investigator, the participant or legal guardian is capable of understanding and complying with protocol requirements.

Exclusion Criteria:

1. Has any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
2. Has received any investigational compound within 30 days (or 5 half- lives of the compound, if longer) before check-in (Day -1).
3. Has received TAK-385 in a previous clinical study.
4. Has current or recent (within 6 months) history of gastrointestinal disease that would be expected to influence the absorption of drugs (ie, history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent heartburn, or any surgical intervention).
5. Is lactose intolerant.
6. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 4 alcoholic drinks per day) within 1 year before screening or is unwilling to agree to abstain from alcohol and drugs throughout the study.
7. Has a positive test result for hepatitis B surface antigen (HBsAG) or hepatitis C virus (HCV) antibody at Screening.
8. Has a positive urine drug result for drugs of abuse or alcohol at Screening or check-in (Day -1).
9. Has taken any prescription medicine or herbal preparations (eg, St. John's wort) or received any immunizations within 30 days before check-in (Day -1).
10. Has taken any OTC medications or vitamin supplements within 14 days before check-in (Day -1). Excluded from this list is occasional use of acetaminophen (paracetamol) ≤ 1 g/day or other medication approved by the sponsor on a case-by-case basis.
11. Is unwilling to agree to abstain from caffeine and food products from 72 hours before check-in (Day -1) to completion of the study.
12. Has a clinically significant electrocardiogram (ECG) abnormality at Screening or check-in (Day -1) or a QTc interval (by the Fridericia correction) of 450 msec or greater. The participant has a history of cardiac disease including, but not limited to, congenital long-QT syndrome, torsades de pointes or torsades de pointes risk factors (eg, cardiac insufficiency, hypokalemia, family history of long-QT syndrome, current use of Class IA [eg, quinidine or procainamide] or Class III [eg, amiodarone or sotalol] antiarrhythmic medications or other medications with known effects on QT interval).
13. Has abnormal laboratory values suggesting a clinically significant disease at Screening or check-in (Day -1) or has abnormalities in the following laboratory parameters: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) value >1.5 times the upper limit of normal.
14. Has engaged in heavy exercise (marathon running, weight lifting, etc) within 72 hours before check-in (Day -1) or is unwilling to agree to abstain from heavy exercise throughout the study.
15. Has known allergy to TAK-385 or its excipients.
16. Participants who, for any reason, are deemed by the investigator to be inappropriate for this study, including participants who are unable to communicate or to cooperate with the investigator.
17. Any participant who is an immediate family member, investigational site employee, or in a dependent relationship with an investigational site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Tempe, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 02 March 2015 to 11 June 2015.
Pre-assignment Details: Healthy participants were enrolled equally in 1 of 2 treatment arms each with 6 sequences that determined the order of administration of TAK-385 tablet formulations. Arm 1: T2 fasted, T4 B fasted or T4 B fed and Arm 2: T2 fasted, T4 C fasted or T4 C fed.
Period: Period 1
Arm/Group | Arm 1: T2-A + T4B-B + T4B-C | Arm 2: T2-A + T4C-D + T4C-E
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Arm 1: T2-A + T4B-B + T4B-C | Arm 2: T2-A + T4C-D + T4C-E
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Arm 1: T2-A + T4B-B + T4B-C | Arm 2: T2-A + T4C-D + T4C-E
Started | 27 | 27
Completed | 27 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: T2-A + T4B-B + T4B-C | Arm 2: T2-A + T4C-D + T4C-E | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (11.62) | 38.8 (10.08) | 38.9 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 27 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black or African American | 4 | 4 | 8
  Multiple | 0 | 1 | 1
  White | 23 | 21 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 21 | 14 | 35
  Not Hispanic or Latino | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54
Weight [Mean (Standard Deviation); unit: kg] | 83.07 (11.957) | 83.69 (13.678) | 83.38 (12.729)
Height [Mean (Standard Deviation); unit: cm] | 174.3 (10.10) | 175.4 (6.79) | 174.8 (8.54)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.311 (2.7624) | 27.148 (3.6504) | 27.230 (3.2074)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: Pharmacokinetic (PK)-Evaluable population included participants who had sufficient dosing and PK data for analysis, and who did not receive any excluded medications.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Arm 1: T2 Formulation Fasted; Arm 2: T2 Formulation Fasted: T2 Formulation Regimen A (T2-A) TAK-385, 120 mg tablet (80 mg + 40 mg tablets), orally, under fasted conditions, once on the first day of one of the 3 treatment periods (Day 1, Day 11 or Day 21).
- Arm 1: T4 Formulation B Fasted: T4 Formulation B Regimen B (T4B-B) TAK-385, 120 mg tablet, orally, under fasted conditions, once on the first day of one of the 3 treatment periods (Day 1, Day 11 or Day 21).
- Arm 1: T4 Formulation B Fed: T4 Formulation B Regimen C (T4B-C) TAK-385, 120 mg tablet, orally, under fed conditions, once on the first day of one of the 3 treatment periods (Day 1, Day 11 or Day 21).
- Arm 2: T4 Formulation C Fasted: T4 Formulation C Regimen D (T4C-D) TAK-385, 120 mg tablet, orally, under fasted conditions, once on the first day of one of the 3 treatment periods (Day 1, Day 11 or Day 21).
- Arm 2: T4 Formulation C Fed: T4 Formulation C Regimen E (T4C-E) TAK-385, 120 mg tablet, orally, under fed conditions, once on the first day of one of the 3 treatment periods (Day 1, Day 11 or Day 21).
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 27
ng/mL | 46.7 (114.9) | 42.0 (153.1) | 33.0 (115.5) | 52.0 (93.3) | 43.5 (146.8) | 41.2 (105.9)
Statistical Analysis 1: Comparison: Arm 1: T2 Formulation Fasted vs Arm 1: T4 Formulation B Fasted; Test type: Superiority or Other; Geometric Mean Ratio = 87.09, 90% CI 2-sided [58.56 to 129.52] — T4 Formulation B Fasted (test)/T2 Formulation Fasted (reference)*100
Statistical Analysis 2: Comparison: Arm 2: T2 Formulation Fasted vs Arm 2: T4 Formulation C Fasted; Test type: Superiority or Other; Geometric Mean Ratio = 83.09, 90% CI 2-sided [59.95 to 115.18] — T4 Formulation C Fasted (test)/T2 Formulation Fasted (reference) * 100
Statistical Analysis 3: Comparison: Arm 1: T4 Formulation B Fasted vs Arm 1: T4 Formulation B Fed; Test type: Superiority or Other; Geometric Mean Ratio = 78.59, 90% CI 2-sided [52.88 to 116.79] — T4 Formulation B Fed (test)/T4 Formulation B Fasted (reference) * 100
Statistical Analysis 4: Comparison: Arm 2: T4 Formulation C Fasted vs Arm 2: T4 Formulation C Fed; Test type: Superiority or Other; Geometric Mean Ratio = 94.23, 90% CI 2-sided [67.98 to 130.61] — T4 Formulation C Fed (test)/T4 Formulation C Fasted (reference) * 100

2. Primary Outcome: AUC(0-120): Area Under the Plasma Concentration-Time Curve From Time 0 to 120 Hours Postdose for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: PK-Evaluable population included participants who had sufficient dosing and PK data for analysis, and who did not receive any excluded medications.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 27
ng•hr/mL | 447 (64.7) | 440 (83.3) | 350 (65.0) | 532 (55.4) | 415 (85.1) | 386 (52.4)
Statistical Analysis 1: Comparison: Arm 1: T4 Formulation B Fasted vs Arm 2: T2 Formulation Fasted; Test type: Superiority or Other; Geometric Mean Ratio = 94.53, 90% CI 2-sided [74.83 to 119.40] — T4 Formulation B Fasted (test)/T2 Formulation Fasted (Reference) *100
Statistical Analysis 2: Comparison: Arm 2: T2 Formulation Fasted vs Arm 2: T4 Formulation C Fasted; Test type: Superiority or Other; Geometric Mean Ration = 77.99, 90% CI 2-sided [64.29 to 94.61] — T4 Formulation C Fasted (test)/T2 Formulation Fasted (reference) * 100
Statistical Analysis 3: Comparison: Arm 1: T4 Formulation B Fasted vs Arm 1: T4 Formulation B Fed; Test type: Superiority or Other; Geometric Mean Ratio = 81.08, 90% CI 2-sided [64.21 to 102.37] — T4 Formulation B Fed (test)/T4 Formulation B Fasted (reference) * 100
Statistical Analysis 4: Comparison: Arm 2: T4 Formulation C Fasted vs Arm 2: T4 Formulation C Fed; Test type: Superiority or Other; Geometric Mean Ratio = 92.78, 90% CI 2-sided [76.48 to 112.55] — T4 Formulation C Fed (test)/T4 Formulation C Fasted (reference) * 100

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 27
ng*hr/mL | 476 (63.5) | 467 (82.8) | 372 (64.1) | 563 (55.1) | 440 (84.8) | 409 (51.8)
Statistical Analysis 1: Comparison: Arm 1: T2 Formulation Fasted vs Arm 1: T4 Formulation B Fasted; Test type: Superiority or Other; Geometric Mean Ratio = 94.43, 90% CI 2-sided [74.85 to 119.12] — T4 Formulation B Fasted (test)/T2 Formulation Fasted (reference) * 100
Statistical Analysis 2: Comparison: Arm 2: T2 Formulation Fasted vs Arm 2: T4 Formulation C Fasted; Test type: Superiority or Other; Geometric Mean Ratio = 78.09, 90% CI 2-sided [64.53 to 94.51] — T4 Formulation C Fasted (test)/T2 Formulation Fasted (reference) * 100
Statistical Analysis 3: Comparison: Arm 1: T4 Formulation B Fasted vs Arm 1: T4 Formulation B Fed; Test type: Superiority or Other; Geometric Mean Ratio = 81.16, 90% CI 2-sided [64.36 to 102.34] — T4 Formulation B Fed (test)/T4 Formulation B Fasted (reference) * 100
Statistical Analysis 4: Comparison: Arm 2: T4 Formulation C Fasted vs Arm 2: T4 Formulation C Fed; Test type: Superiority or Other; Geometric Mean Ratio = 92.99, 90% CI 2-sided [76.84 to 112.54] — T4 Formulation C Fed (test)/T4 Formulation C Fasted (reference) * 100

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A SAE is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: From Day 1 to 30 days after the last dose of study drug (Up to 51 days total)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
percentage of participants
  AEs | 4 | 7 | 7 | 4 | 4 | 7
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Shifts From Normal at Baseline in Safety Laboratory Values in More Than 1 Participant
Description: Participants with shifts from normal at Baseline in safety laboratory values (Clinical Chemistry, Hematology and Urinalysis) collected throughout study. Low=below normal reference range, Normal=within reference range, High=above normal reference range and Abnormal=outside of normal reference range.
Time Frame: Baseline and Days 4, 10, 14, 20, 24 and 26
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
participants
  Aspartate aminotransferase (AST)_Normal to Low | 2 | 1 | 3 | 1 | 3 | 0
  Chloride_Normal to Low | 2 | 1 | 2 | 3 | 0 | 1
  Creatinine_Normal to High | 0 | 0 | 0 | 0 | 0 | 2
  Sodium_Normal to High | 2 | 2 | 1 | 3 | 1 | 2
  Urate_Normal to Low | 1 | 2 | 1 | 0 | 0 | 0
  Urate_Normal to High | 1 | 0 | 0 | 0 | 0 | 0
  Basophils_Normal to High | 3 | 3 | 3 | 1 | 1 | 3
  Lymphocytes_Normal to High | 2 | 1 | 0 | 1 | 1 | 2
  Monocytes_Normal to High | 0 | 0 | 3 | 0 | 1 | 1
  Absolute Monocytes_Normal to High | 2 | 2 | 1 | 0 | 0 | 0
  Neutrophils_Normal to Low | 2 | 2 | 0 | 1 | 1 | 1
  Absolute neutrophils_Normal to Low | 2 | 2 | 0 | 1 | 1 | 1
  Occult blood_Normal to Abnormal | 2 | 0 | 0 | 0 | 0 | 0
  Specific gravity_Normal to Abnormal | 2 | 0 | 2 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Electrocardiogram (ECG) Parameters Abnormal and Clinically Significant
Description: A 12-lead ECG was administered. The investigator interpreted the ECG using one of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.
Time Frame: Days 1, 11, 21 and 26
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Markedly Abnormal Vital Sign Measurements
Description: The percentage of participants with any markedly abnormal standard vital sign measurements was collected throughout study.
Time Frame: From Day 1 to Day 26
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
hours | 2.01 [0.500 to 6.00] | 3.00 [0.502 to 12.00] | 3.00 [0.500 to 8.00] | 3.00 [0.499 to 6.02] | 3.00 [0.499 to 12.0] | 3.00 [1.00 to 8.00]

9. Secondary Outcome: Terminal Phase Elimination Half-Life (T1/2) for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 27 | 27 | 27 | 27 | 27
hours | 36.3 (4.40) | 36.1 (4.90) | 35.1 (4.11) | 34.9 (4.13) | 35.5 (4.22) | 35.4 (2.97)

10. Secondary Outcome: Oral Clearance (CL/F) for TAK-385
Time Frame: Days 1, 11, and 21 predose and at multiple time points (up to 120 hours) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters (L)/hr
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Number analyzed (Participants) | 27 | 26 | 27 | 27 | 27 | 27
liters (L)/hr | 252 (63.6) | 257 (82.7) | 322 (64.0) | 213 (55.1) | 273 (84.8) | 293 (51.9)

ADVERSE EVENTS:
Time Frame: From Day 1 to 30 days after the last dose of study drug (Up to 51 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Arm 1: T2 Formulation Fasted | Arm 1: T4 Formulation B Fasted | Arm 1: T4 Formulation B Fed | Arm 2: T2 Formulation Fasted | Arm 2: T4 Formulation C Fasted | Arm 2: T4 Formulation C Fed
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27 | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 1/27 | 2/27 | 2/27 | 1/27 | 1/27 | 2/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: T2 Formulation Fasted (N=27) | Arm 1: T4 Formulation B Fasted (N=27) | Arm 1: T4 Formulation B Fed (N=27) | Arm 2: T2 Formulation Fasted (N=27) | Arm 2: T4 Formulation C Fasted (N=27) | Arm 2: T4 Formulation C Fed (N=27)
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.